CLINICAL TRIAL: NCT00032734
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Escalation, Multicenter Study Evaluating the Efficacy and Safety of SR121463B in Patients With Syndrome of Inappropriate Antidiuretic Hormone Secretion.
Brief Title: Efficacy of SR121463B in Patients With Syndrome of Inappropriate Antidiuretic Hormone Secretion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI4488; SR121463; LTS5066; LTS10208
Record Dates: First submitted 2002-03-29; First posted 2002-04-01 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Syndrome of Inappropriate ADH (SIADH) Secretion; Hyponatremia
Keywords: Low Blood Sodium (Hyponatremia); SIADH; Inappropriate ADH Syndrome
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia | interventions — satavaptan

INTERVENTIONS:
Drug: satavaptan (SR121463B)

SUMMARY:
The study is designed to assess the efficacy of an investigational drug called SR121463B (vasopressin receptor antagonist) in the treatment of low levels of sodium in the blood associated with the Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH).

This double blind period study is followed by 2 open label extension studies with flexible doses of satavaptan.

DETAILED DESCRIPTION:
This is a multicenter worldwide study with 32 participating men and women aimed to figure out whether SR121463B is safe and effective in correcting low levels of sodium in blood in subjects with SIADH. The participation in the study lasts up to 34 days. After screening, during the first part of the study (maximum 5 days), the subjects receive either capsules of SR121463B or a matching placebo. During the second part of the study (23 days), subjects receive either capsules of SR121463B or no treatment. The subjects will be assessed by physical examinations, electrocardiograms, blood samplings, and urine collections. Women of childbearing potential must have an approved method of contraception.

ELIGIBILITY:
SIADH of any origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-06; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
serum sodium concentration

SECONDARY OUTCOMES:
safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (4):
- Sanofi-aventis Administrative Office, Diegem, Belgium
- Sanofi-aventis Administrative Office, Paris, France
- Sanofi-aventis Administrative Office, Berlin, Germany
- Sanofi-aventis Administrative Office, Budapest, Hungary

REFERENCES:
- See also: Related Info — http://www.centerwatch.com
- See also: Related Info — http://www.sanofi-aventis.com